CLINICAL TRIAL: NCT01728519
Title: Phase I/IIa Study to Assess the Safety, Immunogenicity and Efficacy of AllerT, a Combination of Peptides Derived From Bet v 1, Administered Via the Subcutaneous or Intradermal Route to Volunteers Allergic to Birch Pollen
Brief Title: Phase I/IIa Clinical Evaluation of AllerT vs Placebo in Subjects Allergic to Birch Pollen
Acronym: AN003
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment was stopped before start of the pollen season
Sponsor: Anergis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AN003
Record Dates: First submitted 2012-11-09; First posted 2012-11-20 (Estimated); Last update posted 2012-11-20 (Estimated); Status verified 2012-11

CONDITIONS: Allergic Rhinitis; Allergy
Keywords: Allergy; Birch Pollen; Immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AllerT SC (Experimental): AllerT subcutaneous injections
  Interventions: Drug: AllerT SC
- Placebo SC (Placebo Comparator): placebo subcutaneous injections
  Interventions: Drug: Placebo SC
- AllerT ID (Experimental): AllerT intra-dermal injections
  Interventions: Drug: AllerT ID
- Placebo ID (Placebo Comparator): placebo intra-dermal injections
  Interventions: Drug: Placebo ID

INTERVENTIONS:
Drug: AllerT SC — AllerT subcutaneous injections on days 1, 7, 14, 21 and 56 - cumulative dose 440 microgram)
  Other Names: AllerT subcutaneous injections
  Arms: AllerT SC
Drug: AllerT ID — AllerT intra-dermal injections on days 1, 7, 14, 21 and 56 - cumulative dose 440 microgram)
  Other Names: Aller T intra-dermal injections
  Arms: AllerT ID
Drug: Placebo SC — Placebo subcutaneous injections on days 1, 7, 14, 21 and 56
  Other Names: Placebo subcutaneous injections
  Arms: Placebo SC
Drug: Placebo ID — Placebo intra-dermal injections on days 1, 7, 14, 21 and 56
  Other Names: Placebo intra-dermal
  Arms: Placebo ID

SUMMARY:
Birch pollen allergic patients are currently treated by subcutaneous injections of pollen extracts either by standard allergen specific immunotherapy (SIT) or ultra-rush immunotherapy. Such treatment is prone to side effects and has to be performed in a hospital environment due to the risk of potential anaphylactic reactions. The aim of this study is to test the new product AllerT expected to show widely reduced side effects. AllerT will be injected via two different routes, subcutaneous versus intradermal. The primary endpoint of the study is the local and systemic safety of repeated injections of the product. Since AllerT should provide patients with a pre-seasonal treatment to decrease seasonal allergic symptoms, we will also evaluate the potential efficacy of the approach using a nasal provocation test (NPT) with birch pollen

DETAILED DESCRIPTION:
In addition to the initial protocol, post hoc evaluations were conducted, after new ethics committee reviews, to assess quality of life during the birch pollen season following the trial (April 2009) and to obtain blood samples for evaluation of immunology markers IgG4 and IgE after the season 2010 (July 2010) and after the season 2012 (July 2012),

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis symptoms during the pollen season preceding the study, confirmed by SPT (prick tests) and/or a positive specific IgE CAP test for birch pollen (class I minimum)
* Positive SPT to Bet v 1 (prick tests), negative SPT to AllerT

Exclusion Criteria:

* received immunotherapy against any allergen within 3 years before the start of the study.
* symptomatic to perennial allergens or active seasonal allergy during the trial.
* non controlled asthma (peak flow lower than 30% of predicted value).
* history of any severe medical condition able to influence the course of the study
* Any confirmed or suspected immunodeficiency condition, including human immunodeficiency virus (HIV) infection and asplenia.
* Subjects under immunosuppressive medication.
* Pregnant or lactating women or women willing or intending to become pregnant during the study.
* Any other significant finding which, in the opinion of the investigator, would increase the risk of having an adverse outcome from participating in this protocol or of dropping out of the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 84 days
  collection of local or systemic allergic reactions and any other adverse events through patient diaries and investigators' interviews during the 8-week treatment period and 4 week post-treatment follow-up (Day 84)

SECONDARY OUTCOMES:
change from baseline in blood levels of specific IgG4 and IgE | after 7, 14, 21, 56 and 84 days and after 16 to 18 months and 40 to 42 months
  blood samples were taken at baseline and at weeks 1, 2, 4 and 8 of the treatment period, 4 weeks later and then in July 2010 and in July 2012
change from baseline in nasal provocation tests | 84 days
  nasal provocation tests with birch pollen extract are assessed before treatment and at visit on day 84 of the trial, 4 weeks after completion of treatment

OTHER OUTCOMES:
Total score of the Mini-RQLQ Quality-of-life questionnaire | 4 weeks during April 2009
  weekly questionnaires are filled in by the subjects during April 2009 at the time of the birch pollen season in the trial center area

CONTACTS AND LOCATIONS:
Overall Officials: Francois Spertini, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Lausanne University Hospital, Lausanne, Switzerland